CLINICAL TRIAL: NCT03745508
Title: Influence of Coffee Consumption on BIA-derived Body Composition Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Pro00085821
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2019-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeinated Coffee (200 mg caffeine) (Active Comparator): ~200 mg of caffeine from instant coffee
  Interventions: Other: Instant Coffee
- Caffeinated Coffee (400 mg caffeine) (Active Comparator): ~400 mg of caffeine from instant coffee
  Interventions: Other: Instant Coffee
- Decaffeinated Coffee (Placebo Comparator): Decaffeinated instant coffee
  Interventions: Other: Instant Coffee

INTERVENTIONS:
Other: Instant Coffee — Instant coffee prepared at different caffeine concentrations

SUMMARY:
Body composition analysis is frequently used in both clinical and research settings for evaluation of nutritional status and follow-up. Bioelectrical impedance analysis (BIA) is one method that has been extensively used to measure body composition. To ensure the reliability of BIA results, several recommendations are proposed in the literature. One of them is to avoid coffee and caffeine prior the test. This instruction is primarily based on the potential diuretic effects of caffeine however few studies evaluated the impact of coffee on fluid balance. Research participants usually have several commitments, especially those enrolled in clinical trials. Simplified and evidence-based instructions can avoid unnecessary restrictions and lead to better participant compliance.

DETAILED DESCRIPTION:
Body composition analysis is frequently used in both clinical and research settings for evaluation of nutritional status and follow-up. Using only anthropometric measures is outdated considering the increasing transition towards an individualized treatment and the recent advances in body composition assessment.

Methods to evaluate body composition in humans are chosen mostly based on compartment of interest, study population and feasibility. Bioelectrical impedance analysis (BIA) is one method that has been extensively used to measure body composition. This method uses an impedance that can penetrates both intra- and extracellular fluids to estimate total body water, fat-free mass and body fat.

To ensure the reliability of BIA results, several recommendations are proposed in the literature. One of them is to avoid coffee and caffeine prior the test. This instruction is primarily based on the potential diuretic effects of caffeine, which mechanisms are not completely understood. However, few studies evaluated the impact of coffee or caffeine (supplement) on fluid balance.

Coffee is a highly consumed beverage worldwide. Coffee is one of the most consumed beverage among adults in Canada, and most of the caffeine consumed by adults comes from this beverage. In addition, coffee bioactive compounds such as methylxanthines can influence BIA results due its diuretic effect. Research participants usually have several commitments, especially those enrolled in clinical trials. Simplified and evidence-based instructions can avoid unnecessary restrictions and lead to better participant compliance. To the best of our knowledge the current study is the first to explore the effect of coffee with two different amounts of caffeine on BIA-derived body composition parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 59 years old;
* Body Mass Index between 18.5 and 29.9 kg/m^2.

Exclusion Criteria:

* Women who are menopausal, postmenopausal, pregnant or lactating;
* Use of certain drugs (i.e. diuretics, steroids, growth hormone) or supplements that affects water balance (i.e. creatine);
* Participants who have certain known medical conditions (i.e. cardiovascular, edema, diabetes, kidney disease, liver disease, chronic obstructive pulmonary disease, cancer);
* Participants with any implantable electronic device (e.g. pacemaker, implanted cardiac defibrillator);
* Participants with hypersensitivity to any of the ingredients of the instant coffee.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Body fat predicted by bioelectrical impedance | up to 1.5 hours
  To determine whether the consumption of coffee affects the predicted values of body fat derived by Bioelectrical Impedance Analysis in healthy adults
Body water predicted by bioelectrical impedance | up to 1.5 hours
  To determine whether the consumption of coffee affects the predicted values of body water derived by Bioelectrical Impedance Analysis in healthy adults

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No